CLINICAL TRIAL: NCT03044561
Title: Effect of Sildenafil Citrate on the Outcome of in Vitro Fertilization After Multiple IVF Failures Attributed to Poor Endometrial Development
Brief Title: Sildenafil Citrate of in Vitro Fertilization After Multiple IVF Failures Attributed to Poor Endometrial Development
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr El-Sayed, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: amr el-sayed 2017
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: IVF Failure
MeSH Terms: interventions — Sildenafil Citrate; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil citrate (Experimental)
  Interventions: Drug: Sildenafil Citrate
- placebo (Placebo Comparator)
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: Sildenafil Citrate — 25 mg orally, 4 times per day for 21 days
  Other Names: Silden 25 mg tablet, EIPICO, Inc, Cairo, Egypt
  Arms: Sildenafil citrate
Drug: matching placebo — orally, 4 times per day for 21 days
  Other Names: placebo
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the effect of sildenafil citrate on endometrial development in women with history of recurrent implantation failure after IVF

DETAILED DESCRIPTION:
sildenafil citrate may increase endometrial thickness in women with recurrent IVF failure attributed to poor endometrial development

ELIGIBILITY:
Inclusion Criteria:

* (1) cases of infertility, older than 20 years of age and not older than 40 years.
* (2) Body mass index (BMI):20-29.
* (3) women have experienced two or more implantation failure attributed to inadequate endometrial development.

Exclusion Criteria:

* (1) Uterine abnormalities (e.g. septate, bicornuate and fibroid uterus, Asherman Syndrome).
* (2) Any contraindication to sildenafil citrate or any of the components of its formulation including:

  * Concurrent use of organic nitrites and nitrates.
  * Severe hepatic impairment.
  * Severe renal impairment.
  * Hypotension.
  * Recent stroke or heart attack.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-08-10 (Estimated)

PRIMARY OUTCOMES:
endometrial thickness measures | 21 days
  we will measure endometrial thickness by US in women with recurrent implantation failure

CONTACTS AND LOCATIONS:
Overall Officials: ahmed khairy, professor, Study Director — Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes